CLINICAL TRIAL: NCT03379688
Title: Patient Data Management System Monitored Outcome After Intensive Care, Organdysfunction and Monitoring
Brief Title: PDMS Outcome After Intensive Care, Organdysfunction and Monitoring
Acronym: PONTOS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, PD Dr. med. Dr. rer. nat., MSC, Charite University, Berlin, Germany
Other Study IDs: PONTOS
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pleural Effusion; Blood Pressure
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: Patients undergoing cardiac surgery at Charité Campus Mitte

SUMMARY:
The objective of the explorative registry study is to investigate outcome parameters in the routine treatment of patients who are monitored after heart surgery for either short or long-term treatment in the intensive care unit for close monitoring of blood pressure.

DETAILED DESCRIPTION:
The close monitoring of patients after cardiac surgery is regarded as standard. However, little is currently known about the influence on patient-related outcome parameters. Recently it has already been shown that intraoperative variability of blood pressure during heart surgery has a postoperative effect on 30-day mortality.

The aim of this retrospective study is to investigate the effects of different hemodynamic measurements and management after cardiac surgery on patient-specific outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

1. In-patients of the Charité Universitätsmedizin Berlin
2. at least 18 years old
3. female or male sex
4. cardiosurgical intervention (OPS 5.35 and 5.36) between 01/06 and 12/13.
5. post-operative monitoring of anesthesiological intensive care unit

Exclusion Criteria:

1. previous cardiosurgical interventions during the same hospital stay.
2. incomplete documentation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients who have undergone cardiac surgery in the period 01/06-12/13 at Campus Mitte in the Charité, approx. 7000 patients.
Sampling Method: Probability Sample
Enrollment: 6909 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure in range | Intensive Care stay, an average of 10 days
  Percentage of RR (Blood Pressure) measurements taken by each patient in the target range as a percentage of the total number of measurements taken by that patient.
Blood pressure over range | Intensive Care stay, an average of 10 days
  Percentage of RR measurements of each patient above the target range in relation to the total of all measurements taken by that patient.
Blood pressure below range | Intensive Care stay, an average of 10 days
  Percentage of RR measurements taken by each patient below the target range in relation to the total number of measurements taken by that patient.

SECONDARY OUTCOMES:
Hospital stay | an average of 13 days
  Length of hospital stay
ICU stay | an average of 5 days
  Intensive care unit length of stay
ICU readmission | an average of 30 days
  Amount of hospital readmissions
Renal insufficiency - 1 | intensive care unit stay, an average of 5 days
  Incidence of renal insufficiency
Renal insufficiency - 2 | intensive care unit stay, an average of 5 days
  dialysis duration
Renal insufficiency - 3 | intensive care unit stay, an average of 5 days
  Urine production
Stroke | hospital length of stay, an average of 13 days
  incidence of strokes
Drainage loss | intensive care unit stay, an average of 5 days
  Amount of postoperative drainage loss
transfusions | hospital length of stay, an average of 13 days
  number of transfusions needed
mortality rate-1 | 90 days
  mortality rate after 90 days
mortality rate-2 | 180 days
  mortality rate after 180 days
Pulse Contour Cardiac Output | intensive care unit stay, an average of 5 days
  data received from Pulse Contour Cardiac Output analyses
mortality rate-3 | 5 years
  mortality rate after 5 years
mortality rate-4 | 1 year
  mortality rate after 1 year
Central venous pressure | intensive care unit stay, an average of 5 days
  central venous pressure on intensive care unit
Pleural effusion | hospital length of stay, an average of 13 days
  In-hospital incidence of pleural effusions postoperatively
Case cost | hospital length of stay, an average of 13 days
  Case cost in Euro

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, MD; PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carl M, Alms A, Braun J, Dongas A, Erb J, Goetz A, Goepfert M, Gogarten W, Grosse J, Heller AR, Heringlake M, Kastrup M, Kroener A, Loer SA, Marggraf G, Markewitz A, Reuter D, Schmitt DV, Schirmer U, Wiesenack C, Zwissler B, Spies C. S3 guidelines for intensive care in cardiac surgery patients: hemodynamic monitoring and cardiocirculary system. Ger Med Sci. 2010 Jun 15;8:Doc12. doi: 10.3205/000101. PMID 20577643
- [Background] Aronson S, Stafford-Smith M, Phillips-Bute B, Shaw A, Gaca J, Newman M; Cardiothoracic Anesthesiology Research Endeavors. Intraoperative systolic blood pressure variability predicts 30-day mortality in aortocoronary bypass surgery patients. Anesthesiology. 2010 Aug;113(2):305-12. doi: 10.1097/ALN.0b013e3181e07ee9. PMID 20571360
- [Background] Aronson S, Dyke CM, Levy JH, Cheung AT, Lumb PD, Avery EG, Hu MY, Newman MF. Does perioperative systolic blood pressure variability predict mortality after cardiac surgery? An exploratory analysis of the ECLIPSE trials. Anesth Analg. 2011 Jul;113(1):19-30. doi: 10.1213/ANE.0b013e31820f9231. Epub 2011 Feb 23. PMID 21346163